CLINICAL TRIAL: NCT06398496
Title: Investigating the Effects of an Exercise Intervention on Gut Bacteria, Mood and Cognition in Individuals With Major Depressive Disorder
Brief Title: The Effects of Exercise on Gut Bacteria, Mood and Cognition in Depression
Acronym: Move4Mood
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APC185
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Depressive Disorder, Major
Keywords: gut bacteria; exercise; cardiorespiratory fitness; negative biases
MeSH Terms: conditions — Depressive Disorder, Major; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants randomized to either a control (usual care only) or exercise (usual care + aerobic exercise) intervention group. 'Usual care' is whatever the participant's current treatment plan is, including pharmacological and psychological treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants allocated to usual care study arm, will continue with their current treatment plan as at study enrollment. This includes any pharmacological treatment they may be receiving, as well as any psychological treatment (i.e., therapy sessions with psychiatrist, psychologist etc.). Participants in usual care group will have the same number of study visits (4 total) across a 12-week period, as the aerobic exercise group.
- Aerobic Exercise + Usual Care (Experimental): Participants allocated to aerobic exercise study arm, will engage in aerobic exercise for 12-weeks. This will occur alongside participants usual care, as determined at study enrollment, including any pharmacological treatment they may be receiving, as well as any psychological treatment (i.e., therapy sessions with psychiatrist, psychologist etc.). Participants in aerobic exercise group will have the same number of study visits (4 total) across a 12-week period, as the usual care group.
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — Aerobic exercise intervention will involve multiple exercise sessions completed (unsupervised) by participants. Exercise programs will be given to participants, matched to their current level of fitness as determined via a maximal cardiorespiratory fitness test, and will be adjusted via progressive overload every 1-2 weeks by an exercise and sports science professional.
  Other Names: exercise; cardio; cardiorespiratory exercise
  Arms: Aerobic Exercise + Usual Care

SUMMARY:
This study aims to investigate the effects of a 12-week aerobic (cardio) exercise intervention in people with Major Depressive Disorder.

Measurements taken before, during, and following the 12-week intervention will include assessments of cognition, cardiorespiratory fitness, stress, mood and emotion, and gut bacteria.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) affects 10% of people globally. Additionally, approximately only half of individuals respond to current psychotherapy treatments, with approximately 30% of individuals classed as treatment resistant to psychopharmacological treatments. Despite the current variety in treatments, the gap in efficacy of current treatments means it is imperative to develop a deeper understanding of MDD, so additional treatment options are available to help those whose current treatment is ineffective. Apart from psychotherapies or combined psychopharmacotherapies, exercise may be beneficial for individuals with MDD.

The microbiota-gut-brain-axis has been implicated in MDD, with gut bacteria relative abundance differences observed between individuals with MDD and healthy controls. Exercise interventions can reduce depressive symptoms in individuals with mild-moderate MDD and may be beneficial to people alongside standard care. Physical activity is also capable of modulating the gut microbiome. However, it remains an open question if lifestyle interventions such as exercise may act through the microbiome to enact positive outcomes in individuals with MDD.

As depression does not affect brain function exclusively, but manifests as a whole-body disorder, the investigators propose that depression is, in part, a disorder of the microbiome-gut-brain-axis. Given that the gut microbiome is capable of driving stress and immune alterations that regulate dysfunctional brain circuitry, contributing to depressive symptomology, including cognitive dysfunction and negative biases. Therefore, the current project will be the first to assess the gut microbiome in MDD, whilst undergoing an exercise intervention in conjunction with monitoring dietary intakes.

To achieve this, a RCT will be conducted with two groups of adults with MDD randomized to either a control (usual/standard care) or exercise intervention (aerobic exercise + usual/standard care). The intervention period will last 12-weeks, with those in the exercise group receiving an aerobic exercise program tailored via progressive overload to get them to meet, and then exceed the national physical activity guidelines (>150min of moderate activity per week) by the 12-week mark. Each group will be assessed pre-, mid-, and post-intervention for depressive symptoms, cognition, negative biases, along with diet information, with mechanistic insights gained from evaluation of gut microbiome composition and function, and gut metabolites in the context of microbiota-gut-brain axis signaling.

Prior to enrollment, participants will be informed about the study via a participant information leaflet, and any participant who provides written informed consent to their participation in the study, will then be screened for eligibility and enrolled if eligible.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent.
* Be between 18 and 59 years of age.
* Be in generally good health as determined by the investigator (excluding Major Depressive Disorder diagnosis).
* Community dwelling with a current diagnosis of Major Depressive Disorder, and current depression episode/symptoms as determined via Beck's depression inventory-II (score 13-31).

Exclusion Criteria:

* Change of pharmacological therapy less than 2 weeks prior to beginning of study (including beginning pharmacological treatment).
* Have a significant acute or chronic coexisting illness [cardiovascular, gastrointestinal (GI) [including functional GI disorders, inflammatory bowel disease, coeliac disease], immunological, psychiatric [to include formal/clinical diagnosis or as determined via participant self-report i.e., bipolar spectrum disorder, schizophrenia, or psychosis, but not anxiety disorder], neurodevelopmental or neurodegenerative disorders, metabolic disorders [to include type I or II diabetes], or any condition which contraindicates, in the investigators judgement, entry to the study (including conditions which may prevent an individual from safely participating in low-to-moderate exercise intensities (57-76% heart rate max [HRmax], rating of perceived exertion [RPE]:9-13 (13))-i.e., cardiorespiratory disease[s]).
* Have a malignant disease or any concomitant end-stage organ disease.
* Having a condition or taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk, or confound the interpretation of the study results; to include anti- inflammatory drugs, corticosteroids, laxatives, enemas, proton-pump inhibitors, antibiotics, or probiotics (within 1 month of starting study), anti-coagulants, thrombocyte-aggregation blocking medication(s) and over-the counter non-steroidal analgesics. Participants should have a wash-out period of four-weeks of the above-mentioned medication to be eligible for participation.
* Individuals who are considered to be poor attendees, in the opinion of the investigator, or unlikely for any reason to be able to comply with the trial.
* Participants must not be currently receiving treatment involving experimental drugs. If the participant has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study.
* Are meeting the national physical activity guidelines (16) (i.e., at least 30 minutes a day of moderate intensity activity, five days a week (or 150 minutes a week), specifically in relation to structured aerobic exercise, as assessed via the international physical activity questionnaire (IPAQ). NB: if guidelines are met from occupational or incidental physical activity, individuals would not meet exclusion criteria.
* Current perimenopause, menopause, or post-menopause, in the case of females.
* Females who are pregnant, planning a pregnancy within duration of the study intervention period, or currently lactating.
* Participants who are not fluent in English or English is not first language.
* Are colour blind.
* Have dyslexia or dyscalculia.
* Are a current habitual daily smoker.
* Regular, illegal drug use.
* Alcohol abuse disorder.
* Acute suicidality or suicide attempt in the past 6 months.
* Current eating disorder (anorexia nervosa, bulimia nervosa, binge eating disorder).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Depression symptom change | Change from baseline at 12-weeks
  Depression symptoms measured via self-report questionnaire (Beck's Depression Inventory-II).
Negative and positive affect change | Change from baseline at 12-weeks
  Negative and positive affect, measured via self-report positive affect negative affect schedule.
Gut microbiota change | Change from baseline at 12-weeks
  Gut microbiota, measured via sequencing of stool samples (including measures of diversity, composition, and function).
Cognitive performance: affective perceptual bias | Change from baseline at 12-weeks
  Emotional bias, measured via Emotional bias task via CANTAB.
Cognitive performance: social cognition | Change from baseline at 12-weeks
  Emotional recognition, measured via Emotional recognition task via CANTAB.

SECONDARY OUTCOMES:
Cardiorespiratory fitness change | Change from baseline at 12-weeks
  Cardiorespiratory fitness, measured via VO2max test.
Cognitive performance: Psychomotor function | Change from baseline at 12-weeks
  Reaction time, simple and multi-choice measured via CANTAB.
Cognitive performance: Attention | Change from baseline at 12-weeks
  Rapid Visual Information Processing, measured via CANTAB.
Cognitive performance: Executive Function | Change from baseline at 12-weeks
  Measured via One Touch stockings of Cambridge task, in CANTAB
Cognitive performance: Executive Function/working memory | Change from baseline at 12-weeks
  Measured via Spatial Working Memory task, in CANTAB
Change in concentration of microbial and host metabolites | Change from baseline at 12-weeks
  Assessed via untargeted metabolomics analysis
Change in levels of inflammatory markers | Change from baseline at 12-weeks
  Assessed via inflammatory markers present in stimulated whole blood (including lipopolysaccharide) and unstimulated whole blood samples.
Change in stress symptoms | Change from baseline at 12-weeks
  Measured via the self-report Perceived Stress Scale (PSS). Scale range is from 0-40, higher number(s) indicate higher level of perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Clarke, PhD, Principal Investigator — University College Cork, APC Microbiome Ireland
Locations (1):
- University College Cork, APC Microbiome Ireland, Cork, Cork County, Ireland

IPD SHARING:
Plan to Share IPD: No